CLINICAL TRIAL: NCT04975594
Title: Statin-Intolerance Registry
Acronym: SIR
Status: Active, not recruiting | Type: Observational
Sponsor: University of Leipzig (Other)
Collaborators: University of Jena (Other); University Hospital Dresden (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Ulrich Laufs, Prof. Dr. med, University of Leipzig
Other Study IDs: SIR-2021/05-UKL
Record Dates: First submitted 2021-06-14; First posted 2021-07-23 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Dyslipidemias
Keywords: Statins; Muscle symptoms; Cardiovascular; Lipid Metabolism Disorders
MeSH Terms: conditions — Dyslipidemias; Lipid Metabolism Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Statin-Intolerance Registry will characterize the patient population suffering from statin-intolerance which is a frequent but incompletely understood patient condition with important clinical implications for atherosclerotic cardiovascular disease (ASCVD) prevention.

Patients will be systematically and prospectively included and followed by the registry.

DETAILED DESCRIPTION:
This non-interventional registry based on routine clinical practice will collect data under real-life conditions. The treatment of patients will not be changed by this study.

Data on patient characteristics and the treatment history will be collected via questionnaires at study entree. Yearly follow up visits will re-assess the baseline parameters and document cardiovascular events.

The data will be analyzed using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with dyslipidemia and statin intolerance, defined as:

   Use of 2 or more statins and intolerance of these drugs in any dose or inability to tolerate dosage increasement beyond a maximum weekly dose of 70 mg atorvastatin, 140 mg Simvastatin, pravastatin, or lovastatin, 35 mg rosuvastatin, 280 mg of Fluvastatin and symptoms improve or disappear when statin is reduced in dosage or discontinued
2. Participants are ≧ 18 years old
3. Written declaration of consent is available
4. The patient is cognitively, linguistically and organizationally capable to meet the study requirements. The possibility of 1 year follow-up is very likely.

Exclusion Criteria:

1. Use of any experimental or investigational drugs within 30 days prior to screening.
2. An employee or contractor of the facility conducting the study, or a family member of the principal investigator, co-Investigator, or sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with statin-intolerance
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of treatment adjustments | 3 years
Change in LDL cholesterol level | 3 years

SECONDARY OUTCOMES:
Change in quality of life | 3 years
  by EQ-5D
Development of muscle symptoms over time that initially lead to discontinuation of statin therapy | 3 years
  based on the "Statin-Associated Muscle Symptom Clinical Index" (SAMS-CI)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Laufs, Study Director — University of Leipzig
Locations (1):
- Uniklinik Leipzig, Leipzig, Saxony, Germany